CLINICAL TRIAL: NCT06228118
Title: Clinical Trail of the Lay User Study and Method Comparison Study of Human Chorionic Gonadotropin (HCG) Test System
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: IHC-3000-LCFA01
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Early Pregnancy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Subjects enrolled in method comparison study only
- Subjects enrolled in both the method comparison study and lay user study

SUMMARY:
This clinical trial consisted of lay user study and method comparison study. Method comparison study: evaluate the clinical performance by comparing the results of new device and FDA cleared device (the comparator) tested on the same sample by professionals.

Lay user study: evaluate the usability of by comparing the results of new device on the same sample tested by professionals and lay user, and by lay users complete the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Method comparison study exclusion criteria

   * Female；
   * 18-55 years of age；
   * Voluntary and sign informed consent form.
2. Lay user study inclusion criteria

   * Female；
   * 18-55 years of age；
   * Voluntary and sign informed consent form；
   * Willingness to perform self-test of investigational device；
   * Have the ability to read English.

Exclusion Criteria:

1. Method comparison study exclusion criteria

   * Use of hCG-containing fertility medications (e.g., Pregnyl, Profasi, Novarel, Ovidrel)；
   * Within 8 weeks of childbirth or abortion；
   * The investigator has reason to believe that it is inappropriate for subjects to participate in the study.
2. Lay user study inclusion criteria

   * Use of hCG-containing fertility medications (e.g., Pregnyl, Profasi, Novarel, Ovidrel)；
   * Within 8 weeks of childbirth or abortion；
   * The investigator has reason to believe that it is inappropriate for subjects to participate in the study；
   * Background in a medical or laboratory testing.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 502 subjects with ages from 18-55 years old were enrolled . Among the 502 total subjects, 369 subjects aged between 18 and 55 years old voluntarily participated in the Lay User Study.
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Comparison results | 30minute
  Compare the test results conducted by professionals using investigational device and the comparator, and the positive percent agreement (PPA=100%), negative percent agreement (NPA=100%) and overall percent agreement (OPA=100%) were calculated.

SECONDARY OUTCOMES:
Evaluate the usability and user comprehension of investigational device | 30minute
  The accuracy rate of the critical task is 100%. The Overall Percent Agreement for investigational device is 100% when conducted by a lay user. The accuracy rate of the each questions in the Knowledge assessment is 100%, and 100% of the Ease of operation assessment chose normal, easy, or very easy.

CONTACTS AND LOCATIONS:
Locations (1):
- First Teaching hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, China